CLINICAL TRIAL: NCT07259928
Title: Open-label, Safety, Tolerability and Proof of Concept Study to Evaluate the Use of ANXV (Recombinant Human Annexin A5 Protein) in the Treatment of Patients With Either Diabetic Retinopathy or Recent Onset Retinal Vein Occlusion
Brief Title: Safety and Proof of Concept Study of ANXV (Annexin A5) in Patients With Diabetic Retinopathy or Retinal Vein Occlusion
Acronym: NEXUS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Annexin Pharmaceuticals AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ANN-008; 1012020 (Other: IRAS)
Record Dates: First submitted 2025-09-16; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Non-Proliferative Diabetic Retinopathy; Retinal Vein Occlusion
Keywords: Annexin A5; ANXV; Retinal Vein Occlusion; Non-Profilerative Diabetic Retinopathy; RVO; NPDR
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NPDR, 4mg, 5 doses (Experimental): ANXV 4mg 30 min infusion
  Interventions: Biological: ANXV
- RVO, 4mg, 5 doses (Experimental): ANXV 4mg 30 min infusion
  Interventions: Biological: ANXV
- NPDR, 6 mg, 5 doses (Experimental): ANXV 6mg 30 min infusion
  Interventions: Biological: ANXV
- RVO, 4 mg, 3 doses (Experimental): ANXV 4mg 30 min infusion
  Interventions: Biological: ANXV

INTERVENTIONS:
Biological: ANXV — Human Recombinant Protein Annexin A5

SUMMARY:
The goal of this clinical trial is to learn about the safety of the investigational medicinal product ANXV. It will also learn about how ANXV works to treat non-proliferative diabetic retinopathy and retinal vein occlusion in adults. The main questions it aims to answer are:

* Is ANXV safe to use?
* Does ANXV improve vision or findings related to vision decrease caused by non-proliferative diabetic retinopathy or retinal vein occlusion?
* Does ANXV lower the number of times participants need to use a rescue medication? Researchers will compare different dose levels of ANXV to see what dose would be be appropriate to test in larger studies.

Participants will:

Take ANXV as a 30 minutes infusion (slow injection) for 5 days. Visit the clinic for checkups and tests at 11 visits during 4 months.

DETAILED DESCRIPTION:
The study is an open label, prospective, dose evaluation study to investigate the safety, tolerability and efficacy in patients with Non-Proliferative Diabetic Retinopathy (NPDR) or Retinal Rein Occlusion with recent onset (within 28 days from symptoms onset or diagnosis (whichever is first) to first treatment).

The study consists of 11 visits, whereof one screening visit, five treatment visits and five follow up visits, during a 4 months period.

Intervention is intravenous infusion (30 minutes) with the investigational medicinal product ANXV, a recombinant Annexin A5 protein. The intended dose levels are 4 mg, 1 mg and 6 mg, daily administration for five days.

Safety will be regularly evaluated by the Medical Monitors on a per need basis, as data become available. In case of safety concerns within one indication subset (NPDR and RVO), a lower dose will be initiated within the concerned indication subset (for each subset, independently).

The following assessments will be performed:

Ocular assessments:

* BCVA
* OCT and OCTA
* ERG
* UWF-retinal imaging
* UWF-FFA
* Ocular examination - Slit Lamp biomicroscopy examination, Intraocular Pressure (IOP), RAPD
* Dilated indirect ophthalmoscopy

Non-ocular assessments:

* Vital signs
* ECG
* Safety labs (blood and urine)
* Study labs (blood)

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this trial, an individual must meet all the following criteria:

1. Must have given written informed consent (signed and dated), and any authorizations required by local law and be able to comply with all study requirements
2. Male or female, ≥18 years of age at the time of informed consent
3. Females should have no childbearing potential according to Clinical Trial Facilitation Group (CTFG) definition.
4. Clear ocular media and adequate pupillary dilation in the Study Eye to permit high quality retinal imaging
5. Willing to refrain from unusually strenuous exercise/activity (for example heavy lifting, weight training, intense aerobics classes etc.) for at least 72 hours prior to study visits

   Additionally, NPDR participants must meet the following criteria to be eligible:
6. Diagnosed with moderately severe or severe non-proliferative Diabetic Retinopathy defined as having a DRSS score of 47 and 53 respectively, and no CI-DMO
7. Found to have an ETDRS BCVA score in the study eye (SE) of ≥69 ETDRS (equivalent to Snellen 6/12 or 20/40)

   Additionally, RVO participants must meet the following criteria to be eligible:
8. Diagnosed with Retinal Vein Occlusion with onset of symptoms within 28 days prior to first administration of ANXV

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this trial:

General:

1. Unwillingness or inability to attend all study visits and/or perform all procedures/tests/examinations, including follow-up, as specified by this protocol, or unwillingness to cooperate fully with the Investigator
2. Any major medical or surgical procedure or trauma within 4 weeks prior to the day of trial intervention Treatment 1 (ANXV administration), or planned major surgery within the duration of the study through Day 120
3. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study
4. Prior exposure to a recombinant Annexin A5 protein
5. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to biologics (for example systemically administered recombinant proteins/peptides; a similar drug class to ANXV)
6. Uncontrolled hypertension (systolic > 180 mmHg or diastolic > 110 mmHg)
7. Current use of any systemically administered anti-angiogenic agent (e.g., bevacizumab, sunitinib, cetuximab, sorafenib, pazopanib) or corticosteroids
8. Diagnosed untreated systemic metastasis malignancy
9. A current systemic infection or inflammation that may require antiviral or antimicrobial therapy that will not be completed prior to Screening Visit, or that in the opinion of the Investigator and with concurrence of the Medical Monitor may either put the participant at risk or may influence the results of the study, or the participant's ability to participate in the study
10. Treatment with another investigational drug, biological agent, or device within 3 months of Screening Visit, or 5 half-lives of investigational agent, whichever is longer or planned participation in an interventional trial from signing Informed Consent Form (ICF) through Day 120
11. History of thromboembolic events or deep venous thrombosis within 3 months of Screening Visit
12. Current use of anticoagulant medication (any medications that might have effect on coagulation, haemostasis, and platelets); low dose aspirin allowed prior to informed consent but must be stopped at the time of consent; may begin again 1 day post Treatment 5 infusion
13. Current daily use of benzodiazepines
14. Clinically significant abnormal coagulation parameters at baseline
15. History of autoimmune disease with anticipated presence of persistent Annexin A5 antibodies, e.g., antiphospholipid syndrome, systemic lupus erythematosus, rheumatoid arthritis, Behcet disease or systemic sclerosis
16. Inherited blood disorder (e.g. sickle cell disease, thalassemia)
17. History of unstable coronary artery disease or cerebrovascular accident within the last 3 months
18. Current known kidney disease or evidence of kidney disease and eGFR below 60 mL/min/1.73m2 at baseline
19. Current drug or alcohol abuse as per the opinion of the Investigator, or current excessive nicotine intake (e.g. ≥ 20 cigarettes/day, or equivalent, as per the opinion of the Investigator)
20. Known history of or positive test for chronic infection that affect the immune system (e.g. hepatitis C (HCV), chronic hepatitis B (HBV) and HIV)
21. Class III obesity (Body Mass Index ≥ 40kg/m2), at the time of informed consent
22. Within 6 months prior to the Screening Visit, use of medications known to be toxic to the retina, lens, or optic nerve (e.g., deferoxamine, chloroquine/hydrochloroquine, chlorpromazine, phenothiazines, tamoxifen, and ethambutol)
23. Known hypersensitivity or allergy to fluorescein (e.g., bronchospasm, rash, etc.) or to any component of the study products or a contraindication to dilation of the pupil or fixed pupils; mild allergies without angio-oedema or treatment need may be acceptable if deemed not to be of clinical significance (including but not limited to allergy to animals or mild seasonal hay fever)

    Either or both eyes:
24. A severe (≥0.9 log, Grade 3+ or worse) Relative Afferent Pupillary Defect (RAPD)
25. An IOP greater than 24 mmHg that is not controlled with medication or surgery at the time of the Screening Visit
26. Recent (6 months) history of, or presence of uveitis, presence of intraocular inflammation (history of blepharitis is not exclusionary), current ocular infection
27. Evidence of neovascularization
28. ETDRS BCVA score in the Fellow eye of ≤54 (equivalent to Snellen 6/24 or 20/80)
29. Ocular disorders/additional eye disease, which in the opinion of the Investigator may confound interpretation of study results, compromise protocol assessments or are likely to require intervention during the study, including, but not limited to, atrophy of the retinal pigment epithelium, sub-retinal fibrosis, organized hard exudate plaque, retinal detachment, macular hole, vitreomacular traction, macular epiretinal membrane, clinically significant cataract, vitreous opacities or haemorrhage, glaucoma with documented visual field loss, ischemic optic neuropathy, retinitis pigmentosa or choroidal neovascularization of any cause (e.g., AMD, ocular histoplasmosis, toxoplasmosis, or pathologic myopia)
30. Receipt within the past 6 months or ongoing intravitreal injection of anti-VEGF treatment in either eye

    Study Eye only:
31. Evidence of deep intraretinal haemorrhage involving the centre 1mm of the macula
32. Laser photocoagulation in the study eye within the preceding 6 months prior to the Screening Visit, or likely to receive during the study period
33. Intraocular surgery (including refractive surgery, cataract surgery), or intravitreal (IVT) injection within the preceding 6 months prior to the Screening Visit, or cataract surgery within the preceding 3 months prior to the Screening Visit, or planned intraocular surgery or procedure during the study
34. Recent (6 months) history, or current evidence of ocular herpetic diseases (including herpes simplex virus, varicella zoster or cytomegalovirus)

    NPDR participants will not be eligible if they meet any of the following criteria (only NPDR participants):
35. CI-DMO in either eye which, in the opinion of the Investigator, qualifies for anti-VEGF or laser treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | From day 1 to day 120
  * Incidence and severity of Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
  * Incidence and titre of anti-drug antibodies (ADA) to ANXV pre- and post-administration

SECONDARY OUTCOMES:
Anti-drug antibody | From day 1 to day 120
  Presence of anti-drug antibodies to ANXV
Proof of concept | From day 1 to day 120
  Efficacy measured by eye functional and anatomical assessments.
ANXV concentration | From start of administration up to four hours after start of administration, during all treatment days
  ANXV concentration in blood and urine
Rescue medication use | From day 1 to day 120
  Number of rescue medication occasions

OTHER OUTCOMES:
ANXV binding sites | From day 1 to day 120
  Amount of ANXV binding sites (phosphatidylserine) in plasma and on erythrocytes
Cytokine profile | From day 1 to day 120
  Cytokine profile in plasma
ANXV concentration in urine | Four hours after start of treatment, for the third dose
  ANXV concentration in urine, to evaluate excretion

CONTACTS AND LOCATIONS:
Overall Officials: Anna Frostegård, MD, PhD, Study Director — Annexin Pharmaceuticals AB
Locations (1):
- The Retina Clinic London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD used in a results publication
Supporting Information: Study Protocol, CSR
Time Frame: During the study (as it is an open label study) and during a period after the study that is not yet defined